CLINICAL TRIAL: NCT04308538
Title: Bilateral Lateral Rectus Recession Using Standard Tables Versus Bilateral Lateral Rectus Recession Using Modified Reduced Numbers in Intermittent Exotropia in Children Less Than 6 Years Old
Brief Title: Bil. LR Rec. Using Standard Tables VS Reduced Numbers in Intermittent Exo. in Children Under 6
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Awadein, Prof.Ahmed Awadein, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-20-2020
Record Dates: First submitted 2015-04-18; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Alternating Exotropia
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Recession (Active Comparator): Bilateral lateral rectus muscle recession using standard tables stated by Parks.
  Interventions: Procedure: Standard Recession
- Reduced Recession (Experimental): Bilateral lateral rectus muscle recession using reduced numbers by one millimeter than the standard tables.
  Interventions: Procedure: Reduced Recession

INTERVENTIONS:
Procedure: Standard Recession — Bilateral lateral rectus muscle recession will be performed through fornix approach using standard tables
  Arms: Standard Recession
Procedure: Reduced Recession — Bilateral lateral rectus muscle recession will be performed through fornix approach using reduced numbers
  Arms: Reduced Recession

SUMMARY:
comparing the motor alignment and the incidence of postoperative esotropia following the correction of intermittent exotropia in children below 7 years by bilateral lateral rectus recession using the standard recession tables postulated by Parks versus correction using a reduced recession by one millimeter

ELIGIBILITY:
Inclusion Criteria:

* Patients with poor control intermittent exotropia (where poor control is defined as having a Newcastle score of 3 or more). (9)
* Basic, pseudo- divergence excess and divergence excess types are included.
* If associated with amblyopia it should be corrected before the surgical correction (where the visual acuity will be assessed by the single crowded HOTV test using a commercial projector).

Exclusion Criteria:

* Intermittent exotropia of the convergence insufficiency type.
* Intermittent exotropia with angle of deviation greater than 50 prism diopters.
* Patients with previous squint surgery.
* Patients with secondary deviation due to a sensory lesion or neurological condition.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Motor success rate | 6 months
  Number of patients with orthophoria (8 PD exophoria to 4 PD esophoria)

SECONDARY OUTCOMES:
Pattern strabismus | 6 months
  Number of patients who develop pattern strabismus

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Elshiaty, MD, Study Chair — Cairo University
Locations (1):
- Faculty of Medicine Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Haggerty H, Richardson S, Hrisos S, Strong NP, Clarke MP. The Newcastle Control Score: a new method of grading the severity of intermittent distance exotropia. Br J Ophthalmol. 2004 Feb;88(2):233-5. doi: 10.1136/bjo.2003.027615. PMID 14736781
- [Result] Pratt-Johnson JA, Barlow JM, Tillson G. Early surgery in intermittent exotropia. Am J Ophthalmol. 1977 Nov;84(5):689-94. doi: 10.1016/0002-9394(77)90385-3. No abstract available. PMID 930997
- [Result] Abroms AD, Mohney BG, Rush DP, Parks MM, Tong PY. Timely surgery in intermittent and constant exotropia for superior sensory outcome. Am J Ophthalmol. 2001 Jan;131(1):111-6. doi: 10.1016/s0002-9394(00)00623-1. PMID 11162985
- [Result] Buck D, Powell CJ, Sloper JJ, Taylor R, Tiffin P, Clarke MP; Improving Outcomes in Intermittent Exotropia (IOXT) Study group. Surgical intervention in childhood intermittent exotropia: current practice and clinical outcomes from an observational cohort study. Br J Ophthalmol. 2012 Oct;96(10):1291-5. doi: 10.1136/bjophthalmol-2012-301981. Epub 2012 Aug 11. PMID 22887975